CLINICAL TRIAL: NCT00585208
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Add-On Ramelteon in Ambulatory Bipolar I Disorder With Clinically Significant Sleep Disturbance
Brief Title: Add-On Ramelteon in Bipolar I Disorder With Clinically Significant Sleep Disturbance
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor terminated study
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Takeda (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-11-06-04
Record Dates: First submitted 2007-12-20; First posted 2008-01-03 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Insomnia; Bipolar Disorder
Keywords: insomnia; sleep disturbance; bipolar disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Bipolar Disorder; Parasomnias | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Active Comparator): Ramelteon - this group receives active drug at a fixed dose of 8mg daily throughout study
  Interventions: Drug: Ramelteon
- Placebo (sugar pill) (Placebo Comparator): placebo (sugar pill) - this arm receive the fake pill, also know as placebo or the sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8mg daily
  Other Names: Rozerem
  Arms: Active drug
Drug: Placebo — matching placebo for ramelteon 8mg daily
  Arms: Placebo (sugar pill)

SUMMARY:
The purpose of this research study is to evaluate the safety and efficacy of ramelteon (Rozerem™) as an add-on treatment for sleep problems in patients with bipolar disorder. This study will determine whether or not the addition of ramelteon to ongoing medication(s) for bipolar disorder is useful in improving sleep.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, single site, 8-week trial of add-on ramelteon in outpatient adults (18-65 years old, inclusive) with lifetime bipolar I disorder, with mild to moderate manic symptoms, and currently experiencing a clinically significant sleep disturbance. Approximately 60 subjects will be screened to obtain 30 subjects who enroll in the 8-week trial. Subjects will be randomized to ramelteon or placebo in a double-blind manner as add-on to current treatment. Any other psychotropic medications that the subject is taking at the initiation of participation in this protocol should be continued unchanged throughout the course of this study, except in instances in which these medications require dose reduction for management of side effects. Efficacy and safety assessments will be performed weekly, and the presence of treatment-emergent adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 to 65 years of age, inclusive.
2. Subjects must have lifetime bipolar I disorder as defined by DSM-IV-TR criteria.
3. Subjects' manic symptoms must be mild to moderate in severity, defined as an YMRS score between 10 and 25.
4. Subjects must be currently experiencing a clinically significant sleep disturbance, defined as a PSQI total score > 5.
5. Subjects must be receiving at least 1 mood stabilizing medication, which may include an atypical antipsychotic (e.g., aripiprazole, clozapine, olanzapine, quetiapine, risperidone, ziprasidone) and/or mood stabilizer/anticonvulsant (e.g, lithium, carbamazepine, valproate/divalproex, lamotrigine, oxcarbazepine) medication for > 1 week prior to baseline. Continued administration of benzodiazepines or sedative-hypnotics will be allowed only if the subject has been receiving the medication for > 2 weeks prior to baseline.
6. Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained.
7. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, barrier methods, intrauterine device) for at least 1 month prior to study entry and throughout the study.

Exclusion Criteria:

1. Subjects who are experiencing clinically significant suicidal or homicidal ideation.
2. Subjects who are currently experiencing psychotic symptoms.
3. Subjects with a current DSM-IV-TR Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV-TR diagnosis of a substance dependence disorder within the past 6 months; or, a lifetime DSM-IV-TR psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
4. Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the investigator.
5. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement for > 3 months.
6. Subjects with a clinically significant abnormality in their pre-study physical exam, vital signs, EKG, or laboratory studies.
7. Subjects who are allergic to or who have demonstrated hypersensitivity to ramelteon.
8. Subjects who are taking medications that interact with ramelteon (e.g., ketoconazole, fluconazole, fluvoxamine, rifampin).
9. Females who are pregnant or nursing.
10. Subjects who have received an experimental drug or used an experimental device within 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
Pittsburgh Insomnia Rating Scale (PIRS) | 8 weeks

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | 8 weeks
Inventory of Depressive Symptoms (IDS) | 8 weeks
Hamilton Anxiety Scale (HAM-A) | 8 weeks
Clinical Global Impressions Scale for Bipolar Disorder (CGI-BP) | 8 weeks
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McElroy, MD, Principal Investigator — The Lindner Center of HOPE
Locations (1):
- The Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Winstanley EL, Martens B, Patel NC, Mori N, Moeller D, McCoy J, Keck PE Jr. A randomized, placebo-controlled study of adjunctive ramelteon in ambulatory bipolar I disorder with manic symptoms and sleep disturbance. Int Clin Psychopharmacol. 2011 Jan;26(1):48-53. doi: 10.1097/YIC.0b013e3283400d35. PMID 20861739